CLINICAL TRIAL: NCT04404985
Title: Endovascular vs Surgical Arteriovenous Fistula Outcomes
Acronym: ESAVFO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alian Al-Balas, Associate Clinical Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F0002
Record Dates: First submitted 2020-05-19; First posted 2020-05-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Dialysis Fistula Creation; Endo-vascular AVFs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical AVFs (Active Comparator): Participants who initiated dialysis with a catheter or have advanced chronic kidney disease ,these patients who an Surgical AVF intervention group that will undergo a routine surgical AVF creation.
  Interventions: Procedure: Surgical AVF
- Endo-vascular AVF (Experimental): Participants who initiated dialysis with a catheter or have advanced chronic kidney disease ,these patients who an endo-vascular AVF intervention group that will undergo a per-cutaneous AVF creation.
  Interventions: Procedure: Endo-vascular AVF

INTERVENTIONS:
Procedure: Surgical AVF — Surgical fistula creation is standard surgical procedures, where a small cut through the skin is made to create a channel directly between a vein and artery .
  The study procedures are standard clinical practice, and not considered an experimental procedure.
  Arms: Surgical AVFs
Procedure: Endo-vascular AVF — Endovascular fistula creation is a minimally invasive procedure used to create a canal between close artery and vein at the forearm. A magnet attached to a catheter is passed over a guidewire into the artery while another magnet passed over the guidewire into the vein. The two magnets are aligned close to each other, then the radiofrequency electrode is released from the venous catheter and energized for 2 seconds, creating a channel between the vein and the artery.
  Arms: Endo-vascular AVF

SUMMARY:
Arteriovenous fistulas (AVFs) are the preferred type of vascular access for dialysis, but many of them fail to mature. There are two techniques of creating AVFs either the traditional way with surgery( Surgical AVFs) or novel per-cutaneous technique Endo- AVFs.

Investigators will pilot an randomized clinical trial of endo-AVFs and surgical AVFs at University of Alabama at Birmingham to determine the feasibility of patient recruitment, randomization, and retention. This pilot study will set the stage for a full-scale randomized clinical trial in future.

DETAILED DESCRIPTION:
Arteriovenous fistulas (AVFs) are the preferred type of vascular access for dialysis, but many of them fail to mature. Despite concerted efforts to improve surgical AVF outcomes during the past 20 years, many new AVFs fail to mature, even after interventions to salvage them (assisted maturation). Postoperative ultrasounds of immature AVFs frequently demonstrate decreased flow with narrowing at the anastomosis . Surgically created AVFs typically have a 90o angle at the anastomosis, yet computational fluid dynamics suggest that an anastomotic angle <30o improves the flow hemodynamics. Therefore, there has been great interest in novel AVF technologies to limit vascular injury and improve flow dynamics and maturation rates. The new technology evaluated herein (endovascular AVF (endo-AVF) has the potential to achieve these goals and reduce the cost of vascular access care.

Endo-AVF, a novel per-cutaneous technique of AVF creation, was approved by the FDA in 2018, and has been used in U.S. hemodialysis patients . In contrast to the surgical technique (the current standard), this non-surgical approach (1) minimizes vascular injury at the time of AVF creation and (2) creates a channel between the artery and vein with an angle approaching 0o. These two features provide a scientific rationale for superior maturation compared with that of surgical AVF Investigators will perform a single-center, prospective pilot randomized clinical trial. Investigators will recruit 80 patients who have advanced chronic kidney disease or on hemodialysis with a catheter ,who there pre- operative Ultrasound showed they are eligible to surgical or endo-vascular AVF. Participants will be randomized to one of two groups: an surgical AVF intervention group that will undergo a routine surgical fistula creation, or an endo-vascular AVF intervention group will undergo per-cutaneous fistula creation . Participants will be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Study will include participants who are 18 years and older who are scheduled to have an AVF
* preoperative ultrasound showed feasibility to have an endo-vascular AVF vs surgical upper arm AVF

Exclusion Criteria:

* Age below 18 years
* participants eligible for low forearm AVF ( radio-cephalic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Physiological fistula maturity | 0-6 weeks
  Assess by ultrasound . To assess blood flow within the fistula.
Physiological fistula maturity | 0-6 weeks
  Assess by ultrasound . To assess diameter of the fistula

SECONDARY OUTCOMES:
Clinical fistula maturity | 6 weeks-6 months
  Assess by ultrasound. Able to use the fistula for dialysis
Fistula survival | 0-2 years
  Assess by ultrasound. Continue to able to use fistula for dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No